CLINICAL TRIAL: NCT01619917
Title: The Role of Fractional Vascular Laser Therapy in the Management of Burn Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Sarvesh Logsetty, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B2011: 075
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Burn Scar
Keywords: burn; scar; laser; fractional; vascular
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proximal (Active Comparator): location of the scar proximal to heart
  Interventions: Device: Fractional Vascular Laser
- Distal (Experimental): location of scar distal to heart
  Interventions: Device: Fractional Vascular Laser

INTERVENTIONS:
Device: Fractional Vascular Laser — laser energy will be applied to one of 2 sites (proximal or distal) depending on randomization result

SUMMARY:
While the literature tends to support the use of laser therapy in the management of burn scars, there is a definite lack of appropriately powered, randomized controlled trials. Laser therapy can be quite expensive when compared to other treatment modalities for burn scars, and while promising, its true usefulness has yet to be conclusively demonstrated. For this reason, our assessing the effects of fractional vascular lasers on burn scars. It has been hypothesized that the fractional vascular lasers work on mature scars to decrease scar formation, and the fractional laser works on scar that is quiescent to promote remodelling. The retexturing/ resurfacing of the laser theoretically can decrease the visibility of the mesh pattern created by meshed split thickness skin graft).

Objective:

To determine the benefit of fractional vascular laser treatment in improving burn scar height, texture, vascularity and pliability in late burn scars.

ELIGIBILITY:
Inclusion Criteria:

* living in Winnipeg
* burn scar 6-12 months old
* Fitzpatrick skin type I-III
* thermal burn scar on trunk or extremities

Exclusion Criteria:

* open wound

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2012-11-01; Primary Completion 2027-06-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
reduction in scar appearance | every 3 weeks to 15 weeks
  examine with modified Vancouver Scar Scale

CONTACTS AND LOCATIONS:
Overall Officials: S Logsetty, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada